CLINICAL TRIAL: NCT00017277
Title: A Phase III Double-Blind, Randomized, Placebo-Controlled Study of Erythropoietin When Used as an Adjuvant to Radiation Therapy in Patients With Head and Neck Squamous Cell Carcinoma
Brief Title: Radiation Therapy With or Without Epoetin Alfa in Treating Patients With Head and Neck Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Trans Tasman Radiation Oncology Group (Other); Charite University, Berlin, Germany (Other); Groupe Oncologie Radiotherapie Tete et Cou (Other); Radius Hungaricus Oncology Group (Other); Grup per l'Estudi dels Limfomes de Catalunya i Balears (Other)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: EORTC-22996-24002; EORTC-22996; ARO-EORTC-22996; EORTC-HN-22996; GORTEC-EORTC-22996; TROG-EORTC-22996; RHOG-EORTC-22996; GELCB-EORTC-22996
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Epoetin Alfa; Radiotherapy

INTERVENTIONS:
Biological: epoetin alfa
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Epoetin alfa may help prevent or treat cancer-related anemia. It is not yet known whether radiation therapy is more effective with or without epoetin alfa in treating head and neck cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy with or without epoetin alfa in treating patients who have head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of radiotherapy (in terms of local-regional control) with or without epoetin alfa in patients with squamous cell carcinoma of the head and neck.
* Compare the disease-specific and overall survival of patients treated with these regimens.
* Compare the hemoglobin level of these patients during radiotherapy.
* Compare the acute and late toxic effects of these regimens in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to participating center, site of disease (larynx vs hypopharynx vs oropharynx vs oral cavity), T-classification (T1-2 vs T3-4), N-classification and intent of systematic neck node dissection (N0-1 vs N2-3 without node dissection vs N2-3 with node dissection), hemoglobin level and gender (men with 10-12.5 g/dL vs men with 12.5-14 g/dL vs women with 10-12 g/dL vs women with 12-13.5 g/dL), and type of treatment (EORTC standard vs other vs randomized in other trials). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo standard radiotherapy 5 days a week and receive concurrent epoetin alfa subcutaneously (SC) once weekly.
* Arm II: Patients undergo radiotherapy as in arm I and receive concurrent placebo SC once weekly.

Treatment on both arms continues for 6-8 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed at 3-6 weeks and 9-14 weeks, every 3 months for 2 years, every 6 months for 1 year, and then annually thereafter. After any locoregional recurrence, patients are followed every 6 months for 1 year and then annually thereafter.

PROJECTED ACCRUAL: A total of 800 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the oral cavity, larynx, oropharynx, or hypopharynx

  * Stage T1-T4, any N
  * No T1, N0 glottic tumor
  * No nodal disease from unknown primary
* Previously untreated disease
* No distant metastases
* Planned radiotherapy

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Hemoglobin greater than 10 g/dL but no greater than 14 g/dL for men
* Hemoglobin greater than 10 g/dL but no greater than 13.5 g/dL for women

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No hypertension (diastolic pressure greater than 100 mmHg) refractory to treatment
* No symptomatic cardiovascular disease
* No deep vein thrombosis

Other:

* No other malignancy except cured basal cell skin cancer or carcinoma in situ of the cervix
* No psychological, familial, sociological, or geographical condition that would preclude study compliance
* No smoking during study
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior neoadjuvant chemotherapy
* No concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy to head and neck area
* No concurrent nonconventional radiotherapy

Surgery:

* No prior therapeutic surgery to head and neck area

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2001-03; Primary Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lambin, MD, Study Chair — Maastricht University Medical Center; Jacques Bernier, MD, PhD, Study Chair — Istituto Oncologico della Svizzera Italiana - Ospedale San Giovanni; Jim Denham, MD, Study Chair — Newcastle Mater Misericordiae Hospital; Volker G. Budach, MD, PhD, Study Chair — Charite University, Berlin, Germany; Jean-Henri Bourhis, MD, PhD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris; Ferenc Kaldau, MD, Study Chair — Radius Hungaricus Oncology Group; Anna Sureda, Study Chair — Hospital de la Santa Cruz i Sant Pau
Locations (15):
- Newcastle Mater Misericordiae Hospital, Newcastle, New South Wales, Australia
- Belgium (6):
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - Institut Jules Bordet, Brussels (Bruxelles)
  - Cliniques Universitaires Saint-Luc, Brussels (Bruxelles)
  - Hopital de Jolimont, Haine-Saint-Paul
  - U.Z. Gasthuisberg, Leuven
  - Clinique Sainte Elisabeth, Namur
- Institut Gustave Roussy, Villejuif, France
- Universitaetsklinikum Charite, Berlin, Germany
- Radius Hungaricus Oncology Group, Törökbálint, Hungary
- Rambam Medical Center, Haifa, Israel
- Radiotherapeutisch Instituut Limburg, Heerlen, Netherlands
- Hospital de la Santa Cruz I Sant Pau, Barcelona, Spain
- Ospedale San Giovanni, Bellinzona, Switzerland
- Beatson Oncology Centre, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Result] Bourhis J, Lapeyre M, Tortochaux J, Rives M, Aghili M, Bourdin S, Lesaunier F, Benassi T, Lemanski C, Geoffrois L, Lusinchi A, Verrelle P, Bardet E, Julieron M, Wibault P, Luboinski M, Benhamou E. Phase III randomized trial of very accelerated radiation therapy compared with conventional radiation therapy in squamous cell head and neck cancer: a GORTEC trial. J Clin Oncol. 2006 Jun 20;24(18):2873-8. doi: 10.1200/JCO.2006.08.057. PMID 16782926